CLINICAL TRIAL: NCT04488289
Title: The Föllinge Hypertension and Lifestyle Intervention; a Comparative Study of Methods for Blood Pressure Measurement and Survey of Living Habits
Brief Title: The Föllinge Hypertension and Lifestyle Study
Acronym: FIHST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-01375
Record Dates: First submitted 2020-07-15; First posted 2020-07-27 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Hypertension,Essential; Lifestyle-related Condition
MeSH Terms: conditions — Essential Hypertension; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parallel measurement of blood pressure (Other): Office blood pressure, self-directed and ambulatory blood pressure measurement.
  Interventions: Other: Lifestyle

INTERVENTIONS:
Other: Lifestyle — Cardiovascular risk and lifestyle
  Other Names: Lifestyle intervention

SUMMARY:
Ambulatory blood pressure measurement is more demanding in terms of technical equipment and specially trained staff. If blood pressure measurement in a self-care room is on average equivalent to the ambulatory blood pressure daytime monitoring of hypertension in primary care could be simplified. We therefore want to examine patients monitored for hypertension (ICD 10) with three different methods: conventional blood pressure measurement in office, self-directed automated measurement and ambulatory blood pressure, starting in December 2020. We will also offer an interview covering cardiovascular risk factors, at time for enrollment and after 6 months. The study was approved to include 150 adult study patients (The swedish ethical review authority 2020-01375), men and women, where diagnosis and treatment of hypertension is relevant after a clinical evaluation.

DETAILED DESCRIPTION:
Background: At present, both 24-hour ambulatory blood pressure and self-directed blood pressure measurement in self-care rooms, are services provided by most Swedish primary care clinics. Ambulatory measurement of blood pressure has the disadvantage of being more demanding with regard to the need for advanced technical equipment and trained staff.

Identification of modifiable cardiovascular risk factors and support for change, should be integrated into the treatment programs of hypertension. At study entry all study participants will be invited to an interview focused on identifying modifiable cardiovascular risk factors, with a follow-up interview after six months to consolidate good lifestyle choices.

Aim: If self-directed blood pressure measured in a designated self-care room gives results that are on average equivalent to ambulatory blood pressure daytime, diagnosis and follow-up of hypertensive patients in primary care could be simplified. The majority of patients could then be cared for through self-checks., and the technically more demanding ambulatory blood pressure measurement reserved for special cases. We therefore want to examine patients under treatment or investigated for hypertension in primary care with three different methods: conventional in-office blood pressure measurement by medical staff, ambulatory blood pressure and automated measurement of blood pressure in a special self-care room. Between study entry and after six months changes in modifiable risk factors are documented according to an interview guide covering use of tobacco, alcohol, physical activity and food preferences, with 4-6 fixed alternatives per item.

Demographics: Study patients are recruited among patients registered at Föllinge Health Centre (population 1500), of which about 1000 are in ages where investigation and treatment of hypertension could be relevant. The prevalence of hypertension in the adult population is estimated to about 30%.

Methods: We will recruit men and women from age 20 and older. Advanced age is not a criterion for exclusion if treatment of hypertension is judged to be important after clinical assessment.

Power calculation: Between-methods difference 4 mm Hg, standard deviation 15, correlation 0.4, nominal power 0.8, alpha 0.05: Least necessary number of pairwise measurements N = 135. Corresponding simulation as above, with an assumed correlation 0.5: Necessary number of pairwise measurements N =113. Based on the power calculation, we want to recruit up to 150 study patients for self-directed and office-based blood pressure measurement and ambulatory blood pressure, preliminarily starting in October 1 2020 and last enrolment December 30 2022.

Interview: An interview is offered to all study participants at enrolment and after about 6 months. The interview follows a risk factor inventory according to the Swedish Health Promotion and Healthcare Network, and the patient information pamphlet "Healthy choices make a difference".

Procedures: Potential study patients provide signed informed consent before enrolling in the study. Study patients are identified among patients who are evaluated or treated for hypertension. Study patients who have provided written informed consent are randomised for in-office and self-directed blood pressure measurement in random order on the day before and immediately after completing a 24-hour ambulatory blood pressure measurement.

Technical equipment: Blood pressure measurements are performed with Omron meters (automated oscillometry). In-office: Omron M7 Inteli IT (CE. 01997), certified for arm circumferences 22 - 42 cm. Self-care room: Omron i-Q142 (CE. 0197), certified for arm circumferences 22 - 42 cm. Ambulatory blood pressure measurement: Meditech ABPM-05 Blue BP-05 (CE 0120); cuff width 120 - 250 mm for 23 - 33 cm arm circumference and 150 - 330 mm, for 31 - 40 cm arm circumference.

Office blood pressure: Measurement after five minutes of rest in a quiet environment, with the patient sitting in a chair with a backrest and support for the arms. The blood pressure cuff is applied to the upper arm, at the level of the heart. Three measurements are performed at 1-2 minutes interval. Further measurements are made only if the first two values differ> 10 mm Hg. The blood pressure is recorded as the average of the last two measurements.

Blood pressure in a self-care room: The measurement is performed according to the same principles as in the office. The device signals if the patient does not handle it correctly. Simple instructions are clearly posted in the room. During measurement only one patient may stay in the self-care room at a time, without any staff present. Patients who need supervised instruction are offered guidance before measuring blood pressure on their own.

Ambulatory blood pressure: measurement every 30 minutes from 06 A.M.until 22 P.M. and every 60 minutes at night, for a total of 24 hours. The mean value 06 A.M.- 22 P.M is compared with the mean values for blood pressure measured in-office and in the self-care room respectively. All blood pressure measurements are performed in the left upper arm, to be able to compare with the corresponding values obtained in the self-care room, where the device is adapted for measurement in the left arm, while the patient handles the device's button control with the right hand.

Statistics: Standard numerical outcome measures, means and proportions for baseline variables, t-test and Chi-2, for means and group comparisons, respectively.

Standard blood and urine samples are analysed at the Department of Clinical Chemistry, Östersund Hospital. Potential study patients will undergo a medical examination, relevant biochemical analyses and an ECG recording (12-lead standard ECG) before enrolment in the study.

Importance of expected findings: Ambulatory blood pressure measurement has the disadvantage of being more demanding in terms of technical equipment and specially trained staff. If blood pressure measurement in a self-care room gives results that are equivalent to the ambulatory blood pressure values daytime, monitoring of hypertension in primary care could be simplified.

ELIGIBILITY:
Inclusion Criteria:

* age 20 years or older
* investigated or treated because of essential hypertension
* registered at Föllinge Health Centre

Exclusion Criteria:

* patients in need of emergency care
* advanced stages of disease or dementia
* not able to perform self-directed blood pressure measurement
* pregnancy
* atrial fibrillation
* arm circumference to small or wide for device
* non consenting
* re entry in same study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparative measurement of blood pressure | Hours 24
  Systolic and diastolic pressure, in office, self directed and ambulatory

SECONDARY OUTCOMES:
Assessment of modifiable cardiovascular risk factors | Months 6
  Modifiable risk factor scoring according to the questionnaire "Goda hälsoval gör skillnad" (www.hfsnatverket.se). Higher score indicating higher cardiovascular risk:
  Tobacco, cigarettes per day: never smoker; previous ≥6 months; previous <6 months; daily smoker 1-9; 10-14; 15-20; >20.
  Alcohol, standard glasses per week: abstainer; <1; 1-4; 5-9; 10-14; ≥15 per week. (One standard glass equals 33 cm of beer or cider, 15 cl of wine or 4 cl of spirits.) Binge drinking, standard glasses; men ≥5, women ≥4: Never; <1/month; every month; every week; daily or almost daily.
  Minutes of physic activity for at least 10 minutes, within 1 week: No; <30; 30-60; 60-90; 90-150; 150-300; > 300 minutes (5 hours or more).
  Consumption of vegetables (fresh, boiled or frozen) servings per day: ≥2; 1; 2-6 servings per week; ≤1 servings per week.
  Consumption of fruit (fresh, boiled or frozen) servings per day: ≥2; 1day; 2-6 servings per week; ≤1 servings per week.

CONTACTS AND LOCATIONS:
Locations (1):
- Gunnar Nilsson, Östersund, Region Jämtland Härjedalen, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson G, Lindam A. A comparative trial of blood pressure monitoring in a self-care kiosk, in office, and with ambulatory blood pressure monitoring. BMC Cardiovasc Disord. 2024 Jan 3;24(1):27. doi: 10.1186/s12872-023-03701-1. PMID 38172659